CLINICAL TRIAL: NCT00003010
Title: A Randomized Phase III Trial of Marimastat Versus Placebo in Patients With Metastatic Breast Cancer Who Have Responding or Stable Disease After Induction Chemotherapy
Brief Title: Marimastat or No Further Therapy in Treating Women With Metastatic Breast Cancer That Is Responding or Stable Following Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065585; E2196; NCCTG-E2196
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — marimastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: marimastat

SUMMARY:
RATIONALE: Marimastat may stop the growth of breast cancer by stopping blood flow to the tumor. It is not known whether chemotherapy is more effective with or without marimastat for breast cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of marimastat with that of no further therapy in treating women who have metastatic breast cancer that is responding or stable after chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether marimastat prolongs progression-free survival in women with metastatic breast cancer who have responding or stable disease after receiving standard systemic chemotherapy. II. Determine the toxic effects of marimastat compared with placebo in patients with metastatic breast cancer who have responding or stable disease after receiving standard systemic chemotherapy. III. Determine whether there is an association between trough marimastat concentration and time to disease progression and toxicity.

OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are stratified by the number of involved disease sites at study entry, prior chemotherapy for metastases, osseous disease only at study entry, and bisphosphonate therapy at study entry, and concurrent hormonal therapy (yes vs no). Patients are randomized into two groups. Patients take either marimastat or placebo, one capsule orally twice a day, approximately every 12 hours (i.e., during or after breakfast and dinner). The drug or placebo is given until the development of progressive disease or prohibitive toxicity.

PROJECTED ACCRUAL: A total of 334 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the breast with previous manifestations of progressing regional or metastatic cancer Received one prior systemic chemotherapy regimen for the treatment of metastases, which meets all of the following criteria: Included either doxorubicin, a taxane (i.e., paclitaxel or docetaxel), or both 6-8 courses were given If weekly taxane therapy received, at least 12 doses were given Recovered from all related toxic effects (except alopecia and/or neuropathy) 3-6 weeks have elapsed since last course of chemotherapy was given No more than 40 weeks have elapsed since the first dose of chemotherapy for metastases No current or prior history of brain metastases Responding or stable disease since the initiation of systemic chemotherapy (i.e., no disease progression) required No prior enrollment on ECOG trials for metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal Status: Not specified Performance status: ECOG 0 or 1 Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test required if pre- or peri-menopausal (i.e., last menstrual period within one year prior to study) Pre- or peri-menopausal sexually active women must use effective contraception No other invasive malignancy within last 5 years except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix No history of rheumatoid arthritis, osteoarthritis, symptomatic osteoarthritis requiring therapy, or other inflammatory arthritis At least 5 years since prior invasive malignancies except: Curatively treated basal cell or squamous cell carcinoma of the skin Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No prior trastuzumab Chemotherapy: See Disease Characteristics No concurrent chemotherapy No prior marimastat or batimastat Endocrine therapy: Prior and/or concurrent hormonal therapy for breast cancer allowed Concurrent hormonal therapy allowed Radiotherapy: No concurrent radiotherapy Surgery: No prior organ allograft Other: At least 4 weeks since other investigational agents No concurrent bisphosphonate therapy unless it was initiated prior to the study No concurrent immunosuppressive therapy Patients receiving anticoagulant therapy must be carefully monitored

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 1997-12-02 (Actual); Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Sparano, MD, Study Chair — Albert Einstein College of Medicine; James N. Ingle, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (25):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Zucker S, Wang M, Sparano JA, Gradishar WJ, Ingle JN, Davidson NE; Eastern Cooperative Oncology Group. Plasma matrix metalloproteinases 7 and 9 in patients with metastatic breast cancer treated with marimastat or placebo: Eastern Cooperative Oncology Group trial E2196. Clin Breast Cancer. 2006 Feb;6(6):525-9. doi: 10.3816/cbc.2006.n.006. PMID 16595036
- [Result] Sparano JA, Bernardo P, Stephenson P, Gradishar WJ, Ingle JN, Zucker S, Davidson NE. Randomized phase III trial of marimastat versus placebo in patients with metastatic breast cancer who have responding or stable disease after first-line chemotherapy: Eastern Cooperative Oncology Group trial E2196. J Clin Oncol. 2004 Dec 1;22(23):4683-90. doi: 10.1200/JCO.2004.08.054. PMID 15570070
- [Result] Sparano JA, Bernardo P, Gradishar WJ, et al.: Higher trough marimastat levels are associated with accelerated disease progression and worse survival: results of a randomized phase III trial comparing marimastat with placebo in metastatic breast cancer (MBC) after first-line chemotherapy: an Eastern Cooperative Oncology Group trial (E2196). [Abstract] Breast Cancer Res Treat 76(Suppl 1): A-343, 2002.